CLINICAL TRIAL: NCT03614689
Title: Assessment of the Minimal Residual Disease in Ovarian Cancer From Circulating Tumor DNA and Immune Repertoire
Status: Active, not recruiting | Type: Observational
Sponsor: Geneplus-Beijing Co. Ltd. (Industry)
Collaborators: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RN2017090101
Record Dates: First submitted 2018-07-30; First posted 2018-08-03 (Actual); Last update posted 2024-07-18 (Actual); Status verified 2024-07

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To analyze the proportion of hereditary tumors in ovarian cancer patients in China, as well as the spectrum of variations; the ctDNA characteristics in patients with ovarian cancer; the correlation between the clonal status of mutations and therapy response; whether ctDNA detection can be used to predict the risk of ovarian cancer recurrence; and the characteristics of immune repertoire before and after treatment in patients with ovarian cancer.

DETAILED DESCRIPTION:
100 OC cases with available matched tumor DNA and plasma will be collected. All patients will be treated according to clinical guidelines, and receive circulating tumor DNA (ctDNA) liquid biopsy at the time of diagnosis, at mid treatment, at the end of treatment and during follow-up. The study will be ended when the patients have progressive disease (PD) or reach the longest follow-up time (2 years).

ELIGIBILITY:
Inclusion Criteria:

* Patients who have not received treatment including radiotherapy, chemotherapy, and surgery.
* Expected to achieve satisfactory tumor cytoreductive surgery.
* Estimated lifetime is more than 3 months.
* Understand the research plan and voluntarily participate in the study, sign the informed consent form.
* Ability to collect specimens from each time point and provide corresponding clinical information.

Exclusion Criteria:

* Patients who will receive new adjuvant therapy.
* Patients who have other primary cancer.
* Pregnant or breast-feeding woman.
* Patients with severe mental illness.
* Patients achieve unsatisfactory tumor cytoreductive surgery.
* Patients who voluntarily withdraw for any reason.
* Patients who cannot complete the research plan.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with previously untreated Ovarian Cancer.
Sampling Method: Probability Sample
Enrollment: 104 (Actual)
Dates: Start 2017-11-25 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
The ctDNA characteristics in patients with ovarian cancer , the correlation between the clonal status of mutations and therapy response and whether ctDNA detection can be used to predict the risk of ovarian cancer recurrence. | 2 years

SECONDARY OUTCOMES:
The proportion of hereditary tumors in ovarian cancer patients in China, as well as the spectrum of variations and the characteristics of immune repertoire before and after treatment in patients with ovarian cancer. | 1 years

CONTACTS AND LOCATIONS:
Locations (6):
- China (6):
  - Hunan Cancer Hospital/The Affiliated Cancer Hospital of Xiangya School of Medicine, Central South University, Changsha, Hunan
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi
  - Sichuan Cancer Hospital, Chengdu, Sichuan
  - Affiliated Cancer Hospital of Xinjiang Medical University, Ürümqi, Xinjiang
  - Peking Union Medical College Hospital, Beijing
  - Peking University International Hospital, Beijing